CLINICAL TRIAL: NCT05956015
Title: Albumin Catabolic Rate Measured by a Stable Isotope
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ake Norberg (Other)
Responsible Party: Sponsor-Investigator, Ake Norberg, Associate professor, senior consultant, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2885/2022; K2022-10941 (Other: Karolinska University Hospital)
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Liver Disease Chronic
Keywords: albumin catabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with liver disease (Experimental): patients with chronic liver disease will receive a oral dose of a stable isotope labeled amino acid, 2H5-Phenylalanine, (45 mg/kg body weight 50% MPE).
  Blood samples will be taken over 12 weeks.
  Interventions: Other: stable isotopes
- Healthy volunteers with no signs of liver disease (Experimental): Healthy volunteers with no signs of liver disease will receive a oral dose of a stable isotope labeled amino acid, 2H5-Phenylalanine, (45 mg/kg body weight 50% MPE).
  Blood samples will be taken over 12 weeks.
  Interventions: Other: stable isotopes

INTERVENTIONS:
Other: stable isotopes — The tracer 2H5-phenylalanine is an essential amino acid labeled with deuterium that is a stable isotope, i.e. no radiation is emitted, but the tracer can still be assessed by a combination of gas chromatography and mass spectrometry. The tracer has no measurable effects, but are used for assessment of human physiology.

SUMMARY:
The goal of this physiological study is to compare albumin catabolic rate measured by a stable isotope labeled amino acid in healthy volunteers and in patients with liver disease. At steady state synthesis and catabolism or degradation are equal.

The primary questions it aims to answer are:

* Is albumin catabolic rate lower in patients with liver disease?
* Is albumin catabolic rate measured by stable isotopes in volunteers like historical controls measured by radio-iodinated albumin at the investigator's laboratory or elsewhere? Subjects will be given an oral dose of the deuterium labeled amino acid phenylalanine that will be incorporated by the liver in newly synthetized albumin molecules, and blood samples will be taken over 12 weeks to determine the catabolic rate of albumin.

DETAILED DESCRIPTION:
This study is part of a greater research program investigating the clinical use of albumin infusions in surgery, liver disease and states of critical illness. Indications are still under debate after more than 70 years of use. Good methodology for assessment of synthesis or degradation can be of immense value in these situations.

The gold standard to assess albumin turn-over is to use radio-iodine labeled albumin and take blood samples over several weeks. This method is however associated with many regulatory difficulties and possibly also methodological flaws.

Intravenous injection of deuterium labeled D5-phenylalanine has been used for snap-shot assessment of albumin synthesis, but in this study the stable isotope tracer will be given orally. The idea is that a large dose of labeled phenylalanine will over-flow all body compartments and thus in the liver be incorporated in the newly synthetized albumin molecules. After a short time period there is no more tracer in the amino acid pool and the disappearance of labeled albumin molecules can then be used to measure the albumin disappearance rate, that is equal to the catabolic rate and in steady state also equal to the synthesis rate.

The investigaors believe that by this new method it is possible to overcome some of the issues of radio-iodinated albumin: 1) no radiation, 2) no risk that the tracer leaves from the albumin molecule ahead of the catabolism of the albumin molecule, 3) no risk that the half-life of the albumin molecule is damaged by the labeling process, 4) a potential to measure turn-over of other long-lasting proteins.

Quantitative measurement of enrichment of isotopically labeled phenylalanine is done using gas chromatography-mass spectrometry at the Karolinska Stable Isotope Core where Olav Rooyackers is the laboratory director. Quantification of total phenylalanine (the precursor) is performed by mass spectrometry against an internal standard.

The albumin molecule binds to free acid radicals (scavenger function) with its sulfhydryl group in the Cys-34 position (human mercaptoalbumin). During oxidative stress, the sulfhydryl group is oxidized to sulfinic acid (human non-mercaptoalbumin 1, HNA 1). This is a reversible process. Upon continued oxidation, sulfonic acid is formed, which appears to be irreversible (human non-mercaptoalbumin 2, HNA2). The result is a damaged albumin molecule that has lost its scavenger function. Oxidative stress with high levels of HNA2 may have a decisive role in the pathogenesis of severe liver failure.

There is no data in the literature regarding changes in oxidized albumin over time. The investigators will try to model albumin turnover by looking at how these fractions and the proportions between them change over time. Previous results, suggesting that the amount of oxidized albumin is higher in patients with liver cirrhosis [Oettl 2013], will be reproduced. Finally, the association between albumin oxidation and albumin catabolic rate will be described.

The statistical analysis plan including the determination of the number of study subjects is included in the attached study plan.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

* males and females >= 40 years (to be more like the anticipated age of the liver patients)
* good peripheral blood vessels
* written informed consent

Patients with liver cirrhosis:

* known compensated liver cirrhosis with radiological or endoscopic signs of portal hypertension, such as varices, splenomegaly, or shunts.
* written informed consent

Exclusion Criteria:

* Planned surgical procedure within 3 months (due to possible blood loss i.e. loss of tracer)
* Pregnancy at dosing
* Phenylketonuria
* Participating in other study with stable isotopes within 60 days.
* Circumstance that causes the responsible researcher to assess the research person's participation as inappropriate

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-08-28 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Albumin degradation rate by stable isotope | 12 weeks
  The disappearance rate of 2H5-phenylalanine labeled albumin over time, that is the catabolic rate of albumin, will be measured in both study groups in blood samples over 12 weeks, and the study groups compared.
Albumin degradation rate by different methods | 12 weeks
  Healthy volunteers will be compared to historical controls from our laboratory where albumin degradation rate was measured by radio-iodinated human serum albumin.

SECONDARY OUTCOMES:
Albumin synthesis rate | 120 minutes
  We will compare the oral flooding dose with historical controls where the isotope was given intravenously at our laboratory for measurement of albumin synthesis rates in volunteers and patients with liver disease.
Albumin degradation by modeling different fractions of oxidized albumin over time | 12 weeks
  During the life span of the albumin molecule more and more oxidation appears. The doubly oxidized molecule can no longer reverse to unoxidized albumin. We want to investigate if rations of labeled to unlabeled fractions of the different forms of oxidized albumin can be used for modeling albumin degradation rate
Correlation between oxidation and degradation rate of albumin | 12 weeks
  Oxidation of albumin molecules has been reported to be increased in liver disease. We want to see if there is a correlation between oxidation fraction and albumin degradation rate.

CONTACTS AND LOCATIONS:
Overall Officials: Åke Norberg, PhD, Principal Investigator — Karolinska Institutet, Stockholm
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/15/NCT05956015/Prot_SAP_000.pdf